CLINICAL TRIAL: NCT04585581
Title: Before the Beginning: Preconception Lifestyle Interventions to Improve Future Metabolic Health
Brief Title: Preconception Lifestyle Interventions to Improve Future Metabolic Health (Before the Beginning)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 143756
Record Dates: First submitted 2020-09-25; First posted 2020-10-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Gestational Diabetes
Keywords: Diet therapy; Exercise therapy
MeSH Terms: conditions — Diabetes, Gestational | interventions — High-Intensity Interval Training; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diet + training (Experimental)
  Interventions: Behavioral: time-restricted eating; Behavioral: high intensity exercise; Other: Standard Care
- controls (Active Comparator)
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: time-restricted eating — Participants will be asked to limit the time-window for their daily energy intake to a maximum of 10 hours.
  Arms: diet + training
Behavioral: high intensity exercise — Participants will be encouraged to exercise with high intensity 2-3 times per week
  Arms: diet + training
Other: Standard Care — Standard clinical care

SUMMARY:
The aim of this study is to investigate whether the combination of high intensity exercise and time restricted eating before and during pregnancy can reduce the risk of hyperglycaemia during pregnancy.

DETAILED DESCRIPTION:
Women who are planning a pregnancy will be recruited into a parallel groups randomised controlled trial where the intervention will consist of high intensity training and time-restricted eating. The intervention will continue throughout pregnancy. The investigators will assess whether this lifestyle intervention can effect maternal and offspring cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* contemplating pregnancy within the next six months
* At least one of the following criteria: BMI ≥ 25 < 40 kg/m2, gestational diabetes in a previous pregnancy, previous infant > 4.5 kg, fasting plasma glucose > 5.3 mmol/L, or Non-European ethnicity

Exclusion Criteria:

* On-going pregnancy
* Trying to conceive ≥ 6 cycles at study entry
* Known diabetes (type 1 or 2)
* Shift work that includes night shifts > 2 days per week
* Previous hyperemesis
* Known cardiovascular diseases
* High intensity exercise ≥ 2 hours/week the last 3 months
* Habitual eating window ≤ 12 hours

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose concentration | Gestational week 28
  Plasma glucose concentration after 2 h oral glucose tolerance testing (75 g glucose)

SECONDARY OUTCOMES:
Plasma glucose concentration | Gestational week 12
  Plasma glucose concentration after 2 h oral glucose tolerance testing (75 g glucose)
HbA1c | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Total cholesterol | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Triglycerides | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
High density lipoprotein cholesterol | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Low density lipoprotein cholesterol | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Low density cholesterol | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Glucose | Baseline, intervention week 8, gestational week 12 and 28, and in cord blood (delivery)
  Measured in the blood
Insulin | Baseline, intervention week 8, gestational week 12 and 28, and in cord blood (delivery)
  Measured in the blood
Cytokines | Baseline, intervention week 8, gestational week 12 and 28, and in cord blood (delivery)
  Measured in the blood, a panel of 27 cytokines of relevance for inflammatory status (Bio-Plex Pro Human Cytokine 27-plex Assay)
Adipokines (Adiponectin, Leptin, Ghrelin) | Baseline, intervention week 8, gestational week 12 and 28, and in cord blood (delivery)
  Measured in the maternal blood
Homocysteine | Baseline, intervention week 8, gestational week 12 and 28
  Measured in the maternal blood
Insulin sensitivity | Baseline, intervention week 8, gestational week 12 and 28, and in cord blood (delivery)
  Insulin sensitivity estimated by homeostatic model assessment for insulin resistance (fasting serum insulin concentration (μU/mL) x fasting plasma glucose levels (mmol/L)/22.5)
Total body mass | Baseline, intervention week 8, gestational week 12 and 28
  Estimated using InBody720 bioimpedance scale.
Fat mass | Baseline, intervention week 8, gestational week 12 and 28
  Estimated using InBody720 bioimpedance scale.
Muscle mass | Baseline, intervention week 8, gestational week 12 and 28
  Estimated using InBody720 bioimpedance scale.
Visceral fat area | Baseline, intervention week 8, gestational week 12 and 28
  Estimated using InBody720 bioimpedance scale.
Continuous glucose monitoring | Baseline and 8 weeks intervention
  Continuous glucose monitoring using Freestyle Libre (Abbott Diabetes Care), worn for 14 days.
Cardiorespiratory fitness | Baseline and intervention week 8
  Peak oxygen uptake at a maximum effort exercise test, measured in L/min using Metalyzer.
Blood pressure | Baseline, intervention week 8, gestational week 12 and 28
  Systolic - and diastolic blood pressure (in mmHg) will be measured in the seated position after 15 minutes of rest with an automatic blood pressure device (Welch Allyn, Germany) three times with one minute intervals, in left arm (average of three measurement).
Measured physical activity | Baseline
  Measured by SenseWear activity monitor, worn for 7 days.
Measured physical activity | From baseline and throughout the study period.
  Measured by Amazfit GTS smartwatch
Diet intake | Every 8 week throughout the trial.
  Online food diary (Lifesum app), 4-day registration (one weekend day and three weekdays=
Self-reported physical activity | Baseline, intervention week 8, gestational week 12 and 28, and every 8 week until delivery or until the participant is excluded from the trial due to not conceiving within 6 months from baseline
  International Physical Activity Questionnaire
Sleep | Baseline, intervention week 8, gestational week 12 and 28, and every 8 week until delivery or until the participant is excluded from the trial due to not conceiving within 6 months from baseline
  Self-reported: Pittsburgh Sleep Quality Index
Chronotype | Baseline, intervention week 8, gestational week 12 and 28, and every 8 week until delivery or until the participant is excluded from the trial due to not conceiving within 6 months from baseline
  Self-reported: Hornestberg Morningness Eveningness Questionnaire
Psychological general well being | Baseline, intervention week 8, gestational week 12 and 28, and every 8 week until delivery or until the participant is excluded from the trial due to not conceiving within 6 months from baseline
  Psychological general well being index (PGWBI)
Time to pregnancy | From baseline to pregnancy (up to 36 weeks from enrollment)
  Self-reported
Psychological well-being | Baseline, intervention week 8, gestational week 12 and 28 and every 8 week throughout the trial.
  Self-reported: Psychological General Well Being Index
Birth weight (infant) | Delivery
  From hospital record
Birth length (infant) | Delivery
  From hospital record
Head circumference of infant | Delivery
  From hospital record
Apgar score | Delivery, after 1, 5 and 10 minutes
  From hospital record
ICU admission | Delivery
  From hospital record
Congenital malformation | Delivery
  From hospital record
Gestational age at birth | Delivery
  From hospital record
Length of stay at hospital | Delivery
  From hospital record
Blood pressure (Infant) | Within 72 hours of birth and after 6 weeks post delivery
  Blood pressure (systolic - and diastolic)
Cardiac function (Infant) | Within 72 hours of birth and after 6 weeks post delivery
  Ultrasound echocardiography
  Blood flow and myocardial function will be measured using mechanical wave imaging (MWI).
Infant total body mass | Within 72 hours of birth and after 6 weeks post delivery
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant muscle mass | Within 72 hours of birth and after 6 weeks post delivery
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant fat mass | Within 72 hours of birth and after 6 weeks post delivery
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant hydration status | Within 72 hours of birth and after 6 weeks post delivery
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant bone mass | Within 72 hours of birth and after 6 weeks post delivery
  Estimated using impedance measurements (BioScan tough i8-nano)

OTHER OUTCOMES:
Infant gut microbiome | Within one week of birth, after 6 weeks and after 6 months
  Sequencing of faecal samples
Maternal gut microbiome | After 6 weeks after delivery and after 6 months
  Sequencing of faecal samples
Breastmilk composition | After 6 weeks after delivery and after 6 months
  Breastmilk sampling, for storage (outcomes will be exploratory, not yet specified)
Infant total body mass | At age of 6 months
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant fat mass | At age of 6 months
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant muscle mass | At age of 6 months
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant hydration status | At age of 6 months
  Estimated using impedance measurements (BioScan tough i8-nano)
Infant bone mass | At age of 6 months
  Estimated using impedance measurements (BioScan tough i8-nano)

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology, Fac MH ISB; Kjell Å Salvesen, md prof, Study Director — St Olavs Hospital, Dept Obstetrics & Gynecology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data that underlie the results in publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately following publication, with no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposals, or for individual participant data meta-analyses. Proposals should be directed to trine.moholdt@ntnu.no. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Sujan MJ, Skarstad HM, Rosvold G, Fougner SL, Follestad T, Salvesen KA, Moholdt T. Time restricted eating and exercise training before and during pregnancy for people with increased risk of gestational diabetes: single centre randomised controlled trial (BEFORE THE BEGINNING). BMJ. 2025 Sep 9;390:e083398. doi: 10.1136/bmj-2024-083398. PMID 40925657
- [Derived] Sujan MAJ, Skarstad HMS, Rosvold G, Fougner SL, Nyrnes SA, Iversen AC, Follestad T, Salvesen KA, Moholdt T. Randomised controlled trial of preconception lifestyle intervention on maternal and offspring health in people with increased risk of gestational diabetes: study protocol for the BEFORE THE BEGINNING trial. BMJ Open. 2023 Oct 4;13(10):e073572. doi: 10.1136/bmjopen-2023-073572. PMID 37793933